CLINICAL TRIAL: NCT03504124
Title: Implementing a Multicomponent Intervention to Improve Hypertension Control in Central America
Brief Title: Multicomponent Intervention to Improve Hypertension Control in Central America
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Nutrition of Central America and Panama (Other)
Collaborators: Tulane University School of Public Health and Tropical Medicine (Other); Institute for Clinical Effectiveness and Health Policy (Other); Colorado School of Public Health (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Manuel Ramirez-Zea, Head, INCAP Research Center for the Prevention of Chronic Diseases, Institute of Nutrition of Central America and Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01HL138647-01 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A cluster randomized trial including 32 rural health districts managed by the Ministry of Health (MOH) of Guatemala. Sixteen health districts will be assigned to a multicomponent intervention and 16 to usual care. Each health district will recruit 55 patients aged ≥40 years with uncontrolled hypertension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will receive a multicomponent intervention.
  Interventions: Other: Multicomponent intervention
- Control group (No Intervention): Patients will receive the usual care.

INTERVENTIONS:
Other: Multicomponent intervention — An 18-month multicomponent intervention, which includes protocol-based treatment using: a standard blood pressure (BP) management algorithm, team-based collaborative care, BP audit and feedback, home BP monitoring, and health coaching on antihypertensive medication adherence and lifestyle modification.
  Arms: Intervention group

SUMMARY:
The investigators propose to assess the needs, barriers, and knowledge gaps of hypertension control programs in the national health care systems of the Central America 4 region LMIC (CA-4: Guatemala, Honduras, El Salvador, and Nicaragua); to conduct a cluster randomized trial to test the effect of a multilevel and multicomponent intervention program leveraging an existing subnational primary healthcare system in Guatemala, on blood pressure (BP) control among hypertensive patients; and to evaluate the adaptability, feasibility, fidelity, and sustainability of implementing the program in the primary health care systems of the CA-4 region. The comprehensive intervention, which includes protocol-based treatment using a standard BP management algorithm, team-based collaborative care, BP audit and feedback, home BP monitoring, and health coaching on antihypertensive medication adherence and lifestyle modification, will last for 18 months. This implementation research study presents high public health impact because it will generate urgently needed data on effective, practical, and sustainable intervention strategies aimed at reducing BP related disease burden in Central America and other low- and middle-income countries.

DETAILED DESCRIPTION:
Despite advances in hypertension prevention and treatment research, its prevalence is high and increasing, while the proportions of hypertensive patients who are aware, treated, and controlled are low, especially in low- and middle-income countries (LMIC). The investigators propose to: assess the needs, barriers, and knowledge gaps of hypertension control programs in the national health care systems of the Central America 4 region LMIC (CA-4: Guatemala, Honduras, El Salvador, and Nicaragua); conduct a cluster randomized trial to test the effect of a multilevel and multicomponent intervention program on blood pressure (BP) control among Guatemalan hypertensive patients; and evaluate the adaptability, feasibility, fidelity, and sustainability of implementing the program in the primary health care systems of the CA-4 region. The investigators will conduct formative research to assess the needs of system-wide intervention programs, barriers and facilitators of BP control strategies, and knowledge gaps about implementation for improving hypertension control in the CA-4 health care systems. The proposed trial will recruit 1,770 study participants from 32 primary care districts (55 patients aged ≥22 years with uncontrolled hypertension/district) within a subnational primary care network managed by the Guatemalan Ministry of Health. Sixteen health districts will be assigned to an 18-month multicomponent intervention, which includes protocol-based treatment using: a standard blood pressure (BP) management algorithm, team-based collaborative care, BP audit and feedback, home BP monitoring, and health coaching on antihypertensive medication adherence and lifestyle modification, and 16 to usual care. BP and other indicators will be measured at baseline and at months 6, 12, and 18. The primary clinical outcome is the difference in the proportion of patients with controlled BP (<140/90 mmHg) between the intervention and control groups at 18 months. The secondary outcome is net change in systolic and diastolic BP from baseline to 18 months. Fidelity of the intervention measured monthly by intensification of treatment by provider-teams (titration or addition of new medications) and adherence to medications in patients will be the primary implementation outcome. Other implementation outcomes will be measured every 6 months. The RE-AIM framework will guide the development, implementation, and assessment of the intervention, which will translate and adapt the Hypertension Control Program in Argentina that has been proven effective and feasible. This project have assembled a multidisciplinary investigative team, which will collaborate with the public primary care network in Guatemala to conduct this implementation research project. The intervention and study outcomes are patient-centered, and patients, MOH provider-teams, and other stakeholders will be engaged at every step of the proposed study. The investigators will disseminate the study findings and promote scale-up of the proven effective intervention program, which will generate urgently needed data on effective, adoptable, and sustainable intervention strategies aimed at reducing BP-related disease burden in CA-4 and other low-income settings.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥40 years with BP >140/90 mmHg at the time of enrollment
* Patients who receive care at government health facilities

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1854 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Proportion of controlled blood pressure | 18 months
  Difference in the proportion of patients with controlled blood pressure (<140/90 mmHg) between the intervention and control groups

SECONDARY OUTCOMES:
Change in systolic blood pressure | 18 months
  Net change in systolic blood pressure from baseline to 18 months
Change in diastolic blood pressure | 18 months
  Net change in diastolic blood pressure from baseline to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of Nutrition of Central America and Panama, Guatemala City, Guatemala

REFERENCES:
- [Derived] Paniagua-Avila A, Shelton RC, Figueroa JC, Guzman AL, Gutierrez L, Hernandez-Galdamez DR, Ramirez JM, Rodriguez J, Irazola V, Ramirez-Zea M, Fort MP. Assessing the implementation of a multi-component hypertension program in a Guatemalan under-resourced dynamic context: an application of the RE-AIM/PRISM extension for sustainability and health equity. Implement Sci Commun. 2024 Mar 15;5(1):23. doi: 10.1186/s43058-024-00560-5. PMID 38491376
- [Derived] Paniagua-Avila A, Shelton RC, Guzman AL, Gutierrez L, Galdamez DH, Ramirez JM, Rodriguez J, Irazola V, Ramirez-Zea M, Fort MP. Assessing the implementation of a multi-component hypertension program in a Guatemalan under-resourced dynamic context: An application of the RE-AIM/PRISM extension for sustainability and health equity. Res Sq [Preprint]. 2023 Jan 17:rs.3.rs-2362741. doi: 10.21203/rs.3.rs-2362741/v1. PMID 36712105
- [Derived] Paniagua-Avila A, Fort MP, Glasgow RE, Gulayin P, Hernandez-Galdamez D, Mansilla K, Palacios E, Peralta AL, Roche D, Rubinstein A, He J, Ramirez-Zea M, Irazola V. Evaluating a multicomponent program to improve hypertension control in Guatemala: study protocol for an effectiveness-implementation cluster randomized trial. Trials. 2020 Jun 9;21(1):509. doi: 10.1186/s13063-020-04345-8. PMID 32517806